CLINICAL TRIAL: NCT05019560
Title: Detection of Responsiveness and Awareness in Old Aged Patients During Laryngoscopy and Intubation Using Isolated Forearm Technique
Brief Title: Awareness in Old Aged Patients During Laryngoscopy and Intubation Using Isolated Forearm Technique
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Raham Hasan Mostafa, MD, Assistant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: R 153 / 2021
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Awareness, Anesthesia; Recall Phenomenon; Inhalation; Gas
Keywords: TIVA; Isoflurane; old age
MeSH Terms: conditions — Intraoperative Awareness; Respiratory Aspiration; Mucopolysaccharidosis IV | interventions — Sevoflurane

STUDY DESIGN:
Intervention Model Description: Interventions: Patients were randomized into either Group A (who received inhalational induction) and Group B (who received total intravenous induction followed by maintenance infusion).
  Main outcome measure: IFT response was recorded at laryngoscopy and intubation to identify awareness at this stressful timepoint.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization was performed using a computer-generated random number table in opaque sealed envelopes with 1:1 allocation ratio by an anesthesiologist not directly involved in the trial or patient care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): In group A:
  * The researcher, who supervised the anesthesia, explained the concept of the study to all patients before induction, and then a tourniquet was placed around the dominant arm of the patients after placing a cotton bandage; to be inflated to 200mmHg or 40 mmHg above the systolic blood pressure of the patient; immediately before administration of the muscle relaxant later on.
  * Patients received inhalation induction using sevoflurane 8% and fentanyl 2 µg/kg was administered intravenously. After loss of consciousness, and BIS value of 50 or less, the tourniquet cuff was inflated then atracurium 0.5 mg/kg was given intravenously and sevoflurane reduced to 2%, then laryngoscopy and intubation were done when action of neuromuscular blocker (NMB) was confirmed by the disappearance of T3,T4. During this time, mask assisted ventilation with 100% oxygen was used to achieve normocapnia
  Interventions: Drug: Sevoflurane
- Group B (Active Comparator): In group B:
  * The researcher, who supervised the anesthesia, explained the concept of the study to all patients before induction, and then a tourniquet was placed around the dominant arm of the patients after placing a cotton bandage; to be inflated to 200mmHg or 40 mmHg above the systolic blood pressure of the patient; immediately before administration of the muscle relaxant later on.
  * In group B: propofol 1.5 mg/kg and fentanyl 2 µg/kg were administered intravenously. After loss of consciousness, and BIS value of 50 or less, the tourniquet cuff was inflated and then atracurium 0.5 mg/kg was given intravenously. Propofol infusion 6 mg/kg/hr was started, until action of neuromuscular blocker (NMB) was confirmed by disappearance of T3,T4, then laryngoscopy and intubation were done. The used dosing regimen is according to previous guidelines [8] [9].No inhalational agent was used. Mask assisted ventilation was used to achieve normocapnia.
  Interventions: Drug: TIVA

INTERVENTIONS:
Drug: Sevoflurane — IFT response, hemodynamics and BIS value were recorded during intubation period. Then the data acquisition was stopped and the isolated forearm cuff deflated. IFT values were noted by two independent observers
  Other Names: Inhalational induction
  Arms: Group A
Drug: TIVA — IFT response, hemodynamics and BIS value were recorded during intubation period. Then the data acquisition was stopped and the isolated forearm cuff deflated. IFT values were noted by two independent observers
  Other Names: Total Intravenous induction
  Arms: Group B

SUMMARY:
Awareness during general anesthesia - that has an incidence between 0.1% and 0.9% of cases and may be more in elderly - remains a concern for anesthesiologists. Awareness experiences range from isolated auditory perceptions to reports of a patient being fully awake, immobilized, and in pain. The isolated forearm technique allows assessment of consciousness of the external world (connected consciousness) through a verbal command to move the hand (of a tourniquet-isolated arm) during intended general anesthesia.

DETAILED DESCRIPTION:
Objective: To compare inhalational induction versus intravenous induction regarding awareness during laryngoscopy and intubation in elderly patients undergoing day case elective surgery.

ELIGIBILITY:
Inclusion Criteria:

* 50 American society of anesthesiologists- Physical status (ASA-PS) I and II patients,
* aged 60 to 80 years,
* 70-80 kg,
* both sexes,
* with intact hearing,
* undergoing elective day case surgery were included in the study.

Exclusion Criteria:

1. Uncooperative patients,
2. Language barrier problems,
3. Psychological disorders,
4. Suspected difficult intubation,
5. History of awareness under anesthesia,
6. History of substance abuse,
7. The inability to have tourniquet on arm for the IFT (e.g., lymphedema or operative site)
8. Neuromuscular disorders.
9. Advanced renal, hepatic, cardiac, respiratory or neurological dysfunction
10. If rapid sequence induction was indicated (not suitable for inhalation induction).

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-09-05 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
IFT response was recorded at laryngoscopy and intubation | 10 minutes
  Score is from zero to 5 Increasing score means increasing risk of awareness especially if >3 The primary outcome was IFT response was recorded at laryngoscopy and intubation to identify awareness at this stressful timepoint.

SECONDARY OUTCOMES:
Bispectral index monitor (BIS) | 40 minutes
  Value from 100 to zero. 100 means fully awake We aim to be with in 40-60 intraoperatively to decrease risk of awareness
  BIS values were recorded at the following timings:
  * Baseline
  * After induction and muscle relaxation,
  * During laryngoscopy,
  * After successful intubation
  * After 20 minutes from skin incision
  * After 40 minutes from skin incision
Modified Brice questionnaire | 24 hours
  2 hours and 24 hours after the end of anesthesia, patients were interviewed regarding the experience of dreaming or recall (of the induction period)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request